CLINICAL TRIAL: NCT04326634
Title: Controlled Exercises Effectiveness in Patients With Sleep Apnea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Gema Serrano-Hernanz, PhD, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Geserher
Record Dates: First submitted 2020-03-19; First posted 2020-03-30 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Apnea, Sleep
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Controlled exercises Group (Experimental)
  Interventions: Other: controlled exercises; Other: non controlled exercises group
- Non controlled exercises Group (Experimental)
  Interventions: Other: controlled exercises; Other: non controlled exercises group

INTERVENTIONS:
Other: controlled exercises — controlled exercises
Other: non controlled exercises group — non controlled exercises

SUMMARY:
The aim is to compare a programme of controlled exercises therapy vs a programme of non controlled exercises therapy in patients with sleep apnea

ELIGIBILITY:
Inclusion Criteria:

* sleep apnea

Exclusion Criteria:

* neurologic disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
awake episodes | immediately after treatment
  number of awake episodes
awake episodes | 3 months
  number of awake episodes

IPD SHARING:
Plan to Share IPD: No